CLINICAL TRIAL: NCT06799624
Title: Prognostic Role of molEcular classiFication in Fertility-sparing treAtment of Endometrial canCEr: PREFACE Study
Brief Title: Prognostic Role of molEcular classiFication in Fertility-sparing treAtment of Endometrial canCEr
Acronym: PREFACE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: int
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-01

CONDITIONS: Uterine Cancer
Keywords: uterine cancer; fertility-sparing; molecular classification
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with endometrial cancer eligible for fertility-sparing treatment: Patients diagnosed with endometrial cancer who meet the criteria for inclusion in a fertility-sparing treatment pathway and for whom molecular classification data is available.
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — Only observation following standard of care (histological diagnosis, molecular classification, progestine therapy)

SUMMARY:
Endometrial cancer, the most common gynecologic malignancy in high-income countries, is increasing among reproductive-age women. While hysterectomy prevents pregnancy, hormonal therapies offer fertility-sparing options for select early-stage cases, with ~80% achieving complete response (CR). Molecular classifications (POLEmut, p53abn, MMRd/MSI-H, NSMP) reveal subtype-specific prognostic differences, with NSMP showing higher CR rates and lower recurrence, while p53abn and MMRd/MSI-H fare worse. Recent studies emphasize molecular profiling's potential to guide personalized fertility-sparing treatments. This study explores the prognostic role of these classifications in treatment outcomes.

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic malignancy in high-income countries, with an increasing incidence among women of reproductive age. In 2024, over 65,000 new cases were diagnosed in the United States alone. The prevalence of endometrial cancer in younger women who desire to preserve their fertility presents a significant clinical challenge. Traditional treatment for endometrial cancer involves hysterectomy, which precludes future pregnancies. However, fertility-sparing treatments, primarily using hormonal therapies, have emerged as a viable option for select patients with low-grade, early-stage endometrial cancer. Despite reported complete response (CR) rates of approximately 80% with fertility-sparing therapy, the outcomes vary significantly among patients. Molecular classifications have revolutionized the understanding of endometrial cancer by identifying four distinct subtypes: POLEmut (ultramutated), p53abn (TP53-mutant), MMRd/MSI-H (mismatch repair deficiency/microsatellite instability-high), and NSMP (no specific molecular profile). These classifications have demonstrated prognostic value in predicting oncologic outcomes in endometrial cancer. For instance, the NSMP subtype is associated with higher CR rates (78.4%) and lower recurrence rates (18.4%), whereas MMRd/MSI-H and p53abn subtypes show significantly poorer outcomes, including lower CR rates (48.8% and 50%, respectively) and higher recurrence rates (42.8% and 33%). However, the role of these molecular subtypes in guiding fertility-sparing treatment remains underexplored.

A recent meta-analysis synthesized data from eight studies involving 363 patients who underwent fertility-sparing treatment for endometrial cancer. This analysis highlighted significant differences in complete response to treatment and in oncologic outcomes among the molecular subtypes, emphasizing the potential utility of molecular classification in personalizing treatment strategies. This study aims to build on these findings by prospectively evaluating the prognostic role of molecular classifications in a well-defined cohort of endometrial cancer patients undergoing fertility-sparing treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-45 years with a hysteroscopic confirmed diagnosis of endometrial cancer (FIGO stage IA without myometrial invasion, grade 1 or grade 2, endometrioid histology).
2. Patients desiring fertility preservation
3. Molecular classification of the tumor using next-generation sequencing (NGS) or Proactive Molecular Risk Classifier for Endometrial Cancer (ProMisE).
4. Adequate pre-treatment imaging (MRI or transvaginal ultrasound) confirming no evidence of myometrial invasion or extrauterine spread.

Exclusion Criteria:

1. Patients with atypical endometrial hyperplasia or intraepithelial neoplasia
2. Individuals with tumor samples of insufficient quantity or inadequate quality were not included in the analysis
3. Non-endometrioid histology.
4. Patients with a history of prior uterine malignancy or current synchronous malignancies.
5. Medical contraindications to hormonal therapy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients with endometrial cancer eligible for fertility-sparing treatment.
Study Population: This is a prospective study enrolling patients with endometrial cancer eligible for fertility-sparing treatment.
  Data of consecutive patients treated from the 21st of January 2025.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Response to fertility sparing treatmetn | 12 months
  To assess the differences in Complete Response (CR), Partial response/stable disease (PR/SD) and progression disease (PD) rates among molecular subtypes (NSMP, POLEmut, p53abn, MMRd/MSI-H) of endometrial cancer in patients undergoing fertility-sparing treatment.
Recurrence | 12 months
  To evaluate the recurrence rates of endometrial cancer among these molecular subtypes following fertility-sparing treatment after a CR

SECONDARY OUTCOMES:
Time to CR response | 12 months
  The number of months elapsed from the start of therapy to achieving a complete response.
Obstetric outcomes | 12 mesi
  After fertility-sparing treatment, we assess outcomes such as pregnancy rate (percentage of individuals achieving pregnancy) and live birth rate (percentage of pregnancies resulting in a live baby) for the cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Michigan, Italy

IPD SHARING:
Plan to Share IPD: Undecided